CLINICAL TRIAL: NCT06093048
Title: Endoscopic Retrograde Cholangiopancreatography In Patients Older Than 65Years Old With Obstructive Jaundice: Efficacy And Outcome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Ezzat Mahmoud, specialist of internal medicine sohag university hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Soh-Med-23-10-07MD
Record Dates: First submitted 2023-10-19; First posted 2023-10-23 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Obstructive Jaundice
MeSH Terms: conditions — Jaundice, Obstructive | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): patients with obstructive jaundice equal or older than 65 years old
  Interventions: Procedure: Endoscopic retrograde cholangiopancreatography
- group B (Active Comparator): patients with obstructive jaundice younger than 65 years old
  Interventions: Procedure: Endoscopic retrograde cholangiopancreatography

INTERVENTIONS:
Procedure: Endoscopic retrograde cholangiopancreatography — saftey and outcome in patients older than 65 years old

SUMMARY:
The incidence of pancreato-biliary disorders ,including malignancy, is increasing in elderly patients. Endoscopic retrograde cholangiopancreatography (ERCP) is a well-known therapeutic tool for these pancreato-biliary disorders.

In general, old age is defined as being more than 65 years of age by the World Health Organization. The increase in the domestic aged population is related to the increasing demand for therapeutic ERCP in elderly patients with pancreato-biliary disorders. Common bile duct stones and cancer account for70 % of all jaundice cases in patients over the age of 65 years . This is related to increasing prevalences of cholelithiasis, choledocholithiasis, and malignancy with advancing age .

Endoscopic Retrograde Cholangiopancreatography(ERCP) represents the gold standard technique for the treatment of biliary or pancreatic tract pathology, and it could be often performed with therapeutic intent by realizing procedures such as insertion of bile duct stents and/or endoscopic sphincterotomy. However, evidence about its safety in the elderly is still controversial.

DETAILED DESCRIPTION:
However, therapeutic ERCP is an invasive procedure and is associated with several complications, such as bleeding, pancreatitis, cholangitis, perforation, and mortality. A higher incidence of periprocedural complications might be expected in elderly patients because of the high prevalence of concomitant medical disorders, such as cardiopulmonary and cerebrovascular diseases, and the poor general condition of this population [8].

Despite many previous reports of the safety and efficacy of ERCP in elderly patients, in real clinical practice, there is concern regarding complications of ERCP performed in patients more than 65years old. Also comparative reports of the efficacy and safety of therapeutic ERCP, especially inpatients over 65 years of age, are limited. To investigate this issue, we will evaluate the clinical outcomes such as the technical success rate, procedure-related complications rate, and anesthesia-related adverse events rate of therapeutic ERCP in a older aged group (over than 65 years of age) and control group (less than 65 years of age) at a single tertiary center.

Aim of the work This study aims to evaluate the outcome and safety of ERCP in patients with obstructive jaundice over than 65 years of age.

ELIGIBILITY:
Inclusion Criteria:

* patients with obstructive jaundice older than 18 years old

Exclusion Criteria:

* patients who refuse consent
* patients under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Pancreatitis | 12 months
  serum amylase and lipase using Mann Whitney test
Cholangitis | 12 months
  Temperature chart and serum bilirubin using Chi-square test

SECONDARY OUTCOMES:
Technical success rate | 12 months
  procedure time and frequency of a second ERCP for complete success.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed E Mahmoud, Specialist, Study Director — Sohag University; Mohamed E Mahmoud, Study Director — Sohag University
Locations (1):
- Sohag university Hospital, Sohag, Egypt

REFERENCES:
- [Background] Zhang ZM, Liu Z, Liu LM, Zhang C, Yu HW, Wan BJ, Deng H, Zhu MW, Liu ZX, Wei WP, Song MM, Zhao Y. Therapeutic experience of 289 elderly patients with biliary diseases. World J Gastroenterol. 2017 Apr 7;23(13):2424-2434. doi: 10.3748/wjg.v23.i13.2424. PMID 28428722
- [Background] Ukkonen M, Siiki A, Antila A, Tyrvainen T, Sand J, Laukkarinen J. Safety and Efficacy of Acute Endoscopic Retrograde Cholangiopancreatography in the Elderly. Dig Dis Sci. 2016 Nov;61(11):3302-3308. doi: 10.1007/s10620-016-4283-2. Epub 2016 Aug 26. PMID 27565508
- [Background] Perisetti A, Goyal H, Sharma N. Clinical safety and outcomes of glucagon use during endoscopic retrograde cholangiopancreatography (ERCP). Endosc Int Open. 2022 Apr 14;10(4):E558-E561. doi: 10.1055/a-1747-3242. eCollection 2022 Apr. PMID 35433228
- [Background] Holt BA. Increased severity of post-endoscopic retrograde cholangiopancreatography complications in the elderly: an issue to be addressed. Dig Endosc. 2014 Jul;26(4):534-5. doi: 10.1111/den.12298. No abstract available. PMID 25040209